CLINICAL TRIAL: NCT00850863
Title: Acute and Chronic Inflammatory Responses Induced by Smoking in Individuals Being Susceptible and Non-Susceptible for Development of COPD: From Specific Disease Phenotyping Towards Novel Therapy (Study 2).
Brief Title: Systemic Inflammation in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Top Institute Pharma (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); GlaxoSmithKline (Industry); Nycomed (Industry)
Responsible Party: Professor Dr. J-W.J Lammers, University Medical Center Utrecht
Other Study IDs: 23437
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Inflammation; Smoking; Susceptibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Smoking; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- A: 20 healthy individuals not susceptible for COPD (age 18-40 years, 0 < pack years > 10, FEV1/FVC >70% , FEV1 >85% predicted)
- B: 30 healthy individuals susceptible for COPD (age 40-75years, pack years >20, FEV1/FVC > 70%, FEV1 > 85% predicted)
- C: 20 healthy individuals very susceptible for COPD (age 18-40 year, 0 < pack years > 10, FEV1/FVC > 70%, FEV1 > 85% predicted)and high prevalance of COPD in smoking family members older than 45 years
- D1: 30 COPD patients with GOLD stage I (age 40-75 years, Pack years > 10, FEV1/FVC ≤ 70%, FEV1 > 80% predicted)
- D2: 30 COPD patients with GOLD stage II (age 40-75 years, Pack years > 10, FEV1/FVC ≤ 70%, FEV1 50-80 predicted)
- D3: 30 COPD patients with GOLD stage III (age 40-75 years, Pack years > 10, FEV1/FVC ≤ 70%, FEV1 30-50% predicted)
- D4: 30 COPD patients with GOLD stage IV (age 40-75 years,Pack years > 10, FEV1/FVC ≤ 70%, FEV1 30% predicted)
- E: 20 healthy individuels very susceptible for COPD ( Age 18-40 years,0 < Pack years > 10, FEV1/FVC >70%, FEV1 > 85% predicted, and one of the smoking family members has severe early onset COPD or mild COPD with very low smoke exposure
- F: 30 COPD patients who are highly susceptible (age > 53 years with Pack years > 10 , FEV1/FVC ≤ 70% and FEV1 < 40% predicted) or (age >18 years with 0 < pack years > 5, FEV1/FVC ≤ 70% and FEV1 < 80% predicted)

SUMMARY:
COPD is ranked number 3 by the WHO list of important diseases worldwide and is the only disease with increasing mortality. The pathogenesis of cigarette smoke-induced COPD is obscure, therefore more insight is needed to design effective anti-inflammatory agents. Recently it has become clear that cigarette smoke-induced inflammation is not only present in the lungs but also in the blood, and that this systemic inflammation has important consequences for the clinical expression of COPD. The investigators hypothesize that healthy individuals who are susceptible to cigarette smoking demonstrate a higher and aberrant systemic inflammatory response to cigarette smoke. This susceptibility is caused by heterogeneous factors and is associated with various polymorphic genes that interact with each other and with the environment.

Objective:

* To study systemic inflammation in individuals who are or are not susceptible to develop COPD.
* To characterize the switch to chronicity of the systemic inflmmatory response in COPD
* To determine whether the type and severity of the systemic inflammation contributes to the clinical outcome of COPD
* To compare between subjects who are or are not susceptible to develop COPD in peripheral blood, the corticosteroid responsiveness in vitro, and to unravel underlying mechanisms.
* To study the role of candidate genes that may play a role in the development of fixed airway obstruction, and to identify clues for patient's responsiveness to specific drugs
* To develop new biological and clinical markers for the early diagnosis and monitoring of COPD
* To define possible mediators involved in the early induction of COPD in susceptible smokers, and to define new drug targets

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 and ≤75 years

* Age, pack years, FEV1/FVC and FEV1% predicted must fit in one of the 9 groups of the study population
* Physically and mentally able to undergo the total study protocol
* Written informed consent

Exclusion Criteria:

* Participation in another study
* Alpha-1-antitrypsin deficiency
* Selected grade 1-3 co-morbidity listed in the ACE-27
* Active pulmonary infection like tuberculosis, pneumonia, flue, tracheobronchitis
* Active extra-pulmonary infection like hepatitis A-C, cystitis, gastro-enteritis etc
* Pulmonary diseases like sarcoidosis, pulmonary fibrosis, silicosis, hypersensitivity pneumonitis, asthma
* Life threatening diseases like carcinoma, AIDS (including HIV+), acute leukaemia etc
* Medication that may affect the results of the study: NSAID's, immunosuppressive agents like prednisolon, metotrexate, azathioprine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuels and COPD patients. For detail description see Groups/Cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Systemic inflammation assessed by measurement of expression of established and newly developed markers on innate immune cells; genomic and proteomic analysis of innate immune cells and measurement of pro- and anti-inflammatory cytokines in plasma/serum | 4 years

SECONDARY OUTCOMES:
Extensive clinical characterisation of: a) young healthy individuals with low number of pack years who have a high and low familial risk to develop COPD; b) older individuals with higher number of pack years with either a normal lung function or COPD. | 4 years
Important clinical endpoints include symptoms, lung function, Bode-index, CT-scanning of the lung. | 4 years
Distribution of candidate genes (SNPs) for COPD between the different groups and relations with systemic inflammation. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Lammers, Dr. Prof. MD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Hoonhorst SJ, Lo Tam Loi AT, Pouwels SD, Faiz A, Telenga ED, van den Berge M, Koenderman L, Lammers JW, Boezen HM, van Oosterhout AJ, Lodewijk ME, Timens W, Postma DS, Ten Hacken NH. Advanced glycation endproducts and their receptor in different body compartments in COPD. Respir Res. 2016 Apr 26;17:46. doi: 10.1186/s12931-016-0363-2. PMID 27117828
- [Derived] Hoonhorst SJ, ten Hacken NH, Lo Tam Loi AT, Koenderman L, Lammers JW, Telenga ED, Boezen HM, van den Berge M, Postma DS. Lower corticosteroid skin blanching response is associated with severe COPD. PLoS One. 2014 Mar 12;9(3):e91788. doi: 10.1371/journal.pone.0091788. eCollection 2014. PMID 24622644
- [Derived] Lo Tam Loi AT, Hoonhorst SJ, Franciosi L, Bischoff R, Hoffmann RF, Heijink I, van Oosterhout AJ, Boezen HM, Timens W, Postma DS, Lammers JW, Koenderman L, Ten Hacken NH. Acute and chronic inflammatory responses induced by smoking in individuals susceptible and non-susceptible to development of COPD: from specific disease phenotyping towards novel therapy. Protocol of a cross-sectional study. BMJ Open. 2013 Feb 1;3(2):e002178. doi: 10.1136/bmjopen-2012-002178. Print 2013. PMID 23377993